CLINICAL TRIAL: NCT00459602
Title: A Multi-Center, Laparoscopic Abdominal-Wall Hernia Repair Outcomes Study Using Parietex Composite Mesh
Brief Title: Incisional Hernia Outcomes Study Using Parietex Composite Mesh
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator left institution.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAA7985
Record Dates: First submitted 2007-04-10; First posted 2007-04-12 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Incisional Hernia
Keywords: laparoscopic surgery
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laparoscopic incisional hernia repair: Subjects with an incisional, ventral, umbilical, or spigelian hernia no larger tham 15 cm at the largest measurement, who are candidates for laparoscopic repair of the hernia, and who are able to commit to long-term followup. Laparoscopic repair will proceed as per the standard technique, using polyester mesh.

SUMMARY:
The purpose of this study is to describe the outcomes of laparoscopic incisional hernia repair surgery and to record the outcomes of patients after surgery.

DETAILED DESCRIPTION:
For subjects who agree to participate in this study, participation will last for 1 year. Subjects will undergo all the routine preoperative testing, the same as would be required if they were not participating in this study. This testing includes a blood sample and an electrocardiogram (ECG). Follow up visits will be done at 2 weeks after surgery, 6 weeks after surgery, and 1 year after surgery. Except for the 1 year visit, these office visits are routine and would be requested even if you were not participating in this study. At each of these visits, subjects will be asked about their level of pain and the amount and type of pain medication their are taking. Data gathered for this study will be on outcomes only.

ELIGIBILITY:
Inclusion Criteria:

* incisional hernia suitable for repair by laparoscopic techniques

Exclusion Criteria:

* not a candidate for laparoscopic surgery
* hernia not suitable for laparoscopic repair techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical clinic
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2004-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Visual analog (VAS) scale | 1 year
  pain assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dennis L Fowler, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States